CLINICAL TRIAL: NCT03219814
Title: Does a Cognitive Dissonance-Based Eating Disorder Prevention Intervention Reduce Attentional Biases in Body-Dissatisfied Women?
Brief Title: Cognitive Dissonance and Attentional Biases Related to Body Dissatisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Kristin von Ranson, Associate Professor, Department of Psychology, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REB14-1451
Record Dates: First submitted 2017-07-11; First posted 2017-07-18 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Body-dissatisfaction
Keywords: body-image; attention; cognitive dissonance; eating disorder prevention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be unaware until completion of study as to which group they were assigned to (all participants who sign up are only given the information that they will be engaging in an eyetracking task and discussions about the media). The assessments consist of self-report questionnaires (which will be scores by a masked assessor), and eye-tracking, which is an objective measure of time spent gazing at various stimuli.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cognitive Dissonance Intervention (Experimental): Participants in the Cognitive Dissonance condition will complete tasks from Becker et al.'s (2005) 2-session adaptation of the Body Project. In the intervention groups, participants will be asked to consider the costs of pursuing the thin ideal in verbal, written, and behavioural exercises. Participants will be asked to assume the role as a body activist, and will be given several opportunities to vocalize opposition to the social forces that drive the thin ideal throughout the sessions.
  The first session will involve exercises and discussions about the thin ideal and the costs associated with pursuing it. They will be given a homework assignment to complete at home over the next week. In the following week's session the participants will engage in a role-play exercise, as well as continuing the discussion on the costs of pursuing the thin ideal.
  Interventions: Other: The Body Project
- Mediapsychoeducation Intervention (Active Comparator): Participants in the Mediapsychoeducation condition will complete two sessions of tasks as outlined for Becker et al.'s (2005) media psychoeducation group, which includes no cognitive dissonance tasks. The first session will have the participants discuss the thin ideal and the media's influence on it. They will then watch a 35-minute psychoeducational video on the influence that advertisements have on body image and perpetuating the thin ideal. They will be assigned homework to complete at home during the week between the sessions. The second session will include a discussion surrounding the attainability to the thin ideal, and this discussion will also be expanded to include all forms of media. Participants will then be asked to consider and discuss differences between media images and themselves, as well as whether achieving this "ideal" is realistic, and the costs in trying to achieve this thin ideal. They will then watch a 20-minute video on eating disorders.
  Interventions: Other: Mediapsychoeducation
- Waitlist Control (No Intervention): The participants in the Waitlist condition will be given the Cognitive Dissonance intervention between 5 and 6 weeks after their second assessment-only session (the cognitive dissonance intervention will be offered and scheduled 1 week after their 1-month online follow-up questionnaire).
- Body-Satisfied Assessment Only Condition (No Intervention): Body-satisfied women will be recruited to engage in the assessment portion of the study only (i.e. they will be given NO intervention but are serving as a control in terms of eye-tracking assessment). Body-satisfied women will be assessed to compare their attention to weight words with body-dissatisfied women's attention to weight words. This comparison will be done with an aim of replicating the findings of Tobin (2015), to ensure that for this particular sample, body-dissatisfied women exhibit stronger attentional biases for weight words than body-satisfied women. Attention to weight words in body-satisfied women will be assessed at two time points, one week apart, to ensure there are no spurious changes in attention in body satisfied women.

INTERVENTIONS:
Other: The Body Project — The Body Project is a dissonance-based body-acceptance program designed to help high school girls and college-age women resist cultural pressures to conform to the appearance ideal standard of female beauty and reduce their pursuit of unrealistic bodies. The Body Project is supported by more research than any other body image program and has been found to reduce onset of eating disorders.
  Arms: Cognitive Dissonance Intervention
Other: Mediapsychoeducation — Mediapsychoeducation is used to educate individuals on psychological issues through the use of various medias, in this study mediapsychoeducation is being used to educate individuals on eating disorders and the thin ideal.
  Arms: Mediapsychoeducation Intervention

SUMMARY:
The purpose of this study is to assess a cognitive dissonance-based eating disorder prevention intervention program on its ability to reduce attentional biases in body-dissatisfied women.

DETAILED DESCRIPTION:
Eating disorders are some of the most prevalent psychiatric disorders affecting women in Westernized cultures, and are associated with a range of medical complications; in severe cases, eating disorders can lead to death. Unfortunately, a large proportion of individuals with eating disorders do not receive treatment, and of those who do receive treatment, only approximately 40-50% of clients are symptom-free at the end of treatment. In addition to limited efficacy, existing treatments can be time-consuming and costly. From both public health and humanitarian perspectives it is best to prevent eating disorders prior to their emergence.

This study will use a randomized, controlled design to investigate the effects of a cognitive dissonance-based intervention on attentional biases for weight words in body-dissatisfied women. Cognitive dissonance is thought to occur when there is a discrepancy between one's beliefs or attitudes, and behaviour. The experience of dissonance is thought to create discomfort, and resultantly individuals change their beliefs to be in line with their behaviours. Thus, the core tenet of cognitive dissonance-based interventions is the concept of engaging participants in counter-attitudinal behaviours (e.g., speaking out against the thin ideal) to enact change through cognitive dissonance. This cognitive dissonance-based intervention (The Body Project) targets body dissatisfaction, thin-ideal internalization, and eating disorder symptoms.

Almost all research on the Body Project has assessed its efficacy via self-report, however, this study will use an eye-tracker to measure the gaze. Attentional biases are less susceptible to self-reporting biases than traditional pencil-and-paper questionnaires and so are a more reliable measure of cognitive processing The participants in this study will be placed into one of three different conditions: cognitive dissonance (CD), media psychoeducation (MP), or waitlist control (WL), and a similar number of women will be allocated to the body-satisfied (BS) condition. Both the CD and MP intervention groups will consist of two approximately 2-hour sessions scheduled one week apart, as well as a 30-minute online follow-up questionnaire 1 month after the second intervention/assessment session. Individuals allocated to WL will begin to receive the intervention approximately 5 weeks after the CD and MP groups (after their 1 month follow-up survey). The BS group will consist of two approximately 35- to 40-minute assessment-only sessions scheduled one week apart.

All groups of participants will full out several self-report questionnaire as well as participate in a brief eye-tracking assessment both before and after their allocated intervention group (the BS condition and waitlist control will only complete the questionnaires and eye tracking assessment). Participants will sign up for a group time slot, and the group time slots will be randomly assigned to be given either the CD, and MP, or the WL condition.

Participants will be recruited through the University of Calgary Department of Psychology Research Participation System (RPS) as well as campus community participants recruited through campus advertisements. Potential participants will be pre-screened for the presence of body dissatisfaction (or body satisfaction for the BS assessment only group).

ELIGIBILITY:
Inclusion Criteria:

* body-dissatisfied for three conditions (cognitive dissonance, media psychoeducation, waitlist control)
* body-satisfied for one condition (body-satisfied assessment only condition)
* female-identified for all conditions

Exclusion Criteria:

* male-identified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female identified
Enrollment: 228 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline attentional bias after completing the intervention/control condition, week 2 | change in attentional bias from baseline recorded at the end of the assigned intervention/control condition (week 2)
  using an EyeLink 1000 eye-tracking system gaze will be tracked for biases to view weight words and images

SECONDARY OUTCOMES:
Change from baseline body dissatisfaction after completing the intervention/control condition, week 2 | change in BSQ score from baseline measured at the end of the assigned intervention/control condition (week 2)
  Level of body dissatisfaction will be measured using the Body Shape Questionnaire (BSQ; Cooper, Taylor, Cooper, & Fairburn, 1987).
Change from baseline body dissatisfaction at the one-month follow up | change in BSQ score from baseline measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  Level of body dissatisfaction will be measured using the Body Shape Questionnaire (BSQ; Cooper, Taylor, Cooper, & Fairburn, 1987).
Change from baseline body appreciation after completing the intervention/control condition, week 2 | change in Body Appreciation Scale score measured at the end of the assigned intervention/control condition (week 2)
  body appreciation will be assessed using the the Body Appreciation Scale (Tylka & Wood-Barcalow, 2015).
Change from baseline body appreciation at the one-month follow up | change in Body Appreciation Scale score measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  body appreciation will be assessed using the the Body Appreciation Scale (Tylka & Wood-Barcalow, 2015).
Change from baseline thin-ideal internalization after completing the intervention/control condition, week 2 | change in SATAQ score measured at the end of the assigned intervention/control condition (week 2)
  thin-ideal internalization will be assessed using the internalization subscale of the Sociocultural Attitudes Towards Appearance Questionnaire (SATAQ; Schaefer et al., 2015)
Change from baseline thin-ideal internalization at the one-month follow up | Change in SATAQ score measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  thin-ideal internalization will be assessed using the internalization subscale of the Sociocultural Attitudes Towards Appearance Questionnaire (SATAQ; Schaefer et al., 2015)
Change from baseline eating pathology after completing the intervention/control condition, week 2 | change in EDE-Q score measured at the end of the assigned intervention/control condition (week 2)
  eating pathology will be assessed using the Eating Disorder Examination Questionnaire (EDE-Q 6.0; Fairburn & Beglin, 1994)
Change from baseline eating pathology at the one-month follow up | change in EDE-Q score measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  eating pathology will be assessed using the Eating Disorder Examination Questionnaire (EDE-Q 6.0; Fairburn & Beglin, 1994)
Change from baseline explicit weight stigma after completing the intervention/control condition, week 2 | change in Anti-Fat Attitudes Questionnaire score measured at the end of the assigned intervention/control condition (week 2)
  Explicit weight stigma will be assessed using the Anti-Fat Attitudes Questionnaire (Crandall, 1994)
Change from baseline explicit weight stigma at the one-month follow up | Change in Anti-Fat Attitudes Questionnaire score measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  Explicit weight stigma will be assessed using the Anti-Fat Attitudes Questionnaire (Crandall, 1994)
Change from baseline weight self-stigma after completing the intervention/control condition, week 2 | change in Weight Self-Stigma Questionnaire score measured at the end of the assigned intervention/control condition (week 2)
  Weight self-stigma will be assessed using the Weight Self-Stigma Questionnaire (Lillis et al., 2010)
Change from baseline weight self-stigma at the one-month follow up | change in Weight Self-Stigma Questionnaire score measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  Weight self-stigma will be assessed using the Weight Self-Stigma Questionnaire (Lillis et al., 2010)
Change from baseline state body dissatisfaction after completing the intervention/control condition, week 2 | change in Body Dissatisfaction Visual Analogue Scale score measured at the end of the assigned intervention/control condition (week 2)
  State body dissatisfaction will be assessed using a Visual Analogue Scale that asks participants to rate their current level of body satisfaction/dissatisfaction on a scale from 0 (extremely satisfied with your body) to 100 (extremely dissatisfied with your body)
Change from baseline state body dissatisfaction at the one-month follow up | change in Body Dissatisfaction Visual Analogue Scale score measured in online follow-up survey administered one month after week 2 of the assigned intervention/control condition
  State body dissatisfaction will be assessed using a Visual Analogue Scale that asks participants to rate their current level of body satisfaction/dissatisfaction on a scale from 0 (extremely satisfied with your body) to 100 (extremely dissatisfied with your body)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin von Ranson, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becker, C. B., Smith, L. M., & Ciao, A. C. (2005). Reducing eating disorder risk factors in sorority members: A randomized trial. Behavior Therapy, 36, 245-253. doi:10.1016/S0005-7894(05)80073-5
- [Background] Cooper, P. J., Taylor, M. J., Cooper, Z., & Fairburn, C. G. (1987). The development and validation of the body shape questionnaire. International Journal of Eating Disorders, 6, 485-494. Retrieved from http://search.proquest.com/docview/617439169
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Tylka TL, Wood-Barcalow NL. The Body Appreciation Scale-2: item refinement and psychometric evaluation. Body Image. 2015 Jan;12:53-67. doi: 10.1016/j.bodyim.2014.09.006. Epub 2014 Oct 21. PMID 25462882
- [Background] Van Strien, T., Frijters, J. E., Van Staveren, W. A., Defares, P. B., & Deurenberg, P. (1986). The predictive validity of the Dutch restrained eating scale. International Journal of Eating Disorders, 5(4), 747-755. doi:10.1002/1098-108X(198605)5:4<747::AID-EAT2260050413>3.0.CO;2-6
- [Background] Stice, E., Rohde, P., & Shaw, H. (2013). The Body Project: A dissonance-based eating disorder prevention intervention (Updated ed.). Facilitator guide.
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Crandall CS. Prejudice against fat people: ideology and self-interest. J Pers Soc Psychol. 1994 May;66(5):882-94. doi: 10.1037//0022-3514.66.5.882. PMID 8014833
- [Background] Lillis J, Luoma JB, Levin ME, Hayes SC. Measuring weight self-stigma: the weight self-stigma questionnaire. Obesity (Silver Spring). 2010 May;18(5):971-6. doi: 10.1038/oby.2009.353. Epub 2009 Oct 15. PMID 19834462
- [Derived] Tobin LN, Sears CR, von Ranson KM. Two eating disorder preventive interventions reduce attentional biases in body-dissatisfied university women: A cluster randomized controlled trial. J Consult Clin Psychol. 2022 Dec;90(12):911-924. doi: 10.1037/ccp0000768. Epub 2022 Nov 17. PMID 36395030